# **Study Title**

Predict + Protect: A randomized controlled trial exploring the effectiveness of predictive health education intervention on the adoption of protective behaviors related to influenza-like illness (ILI)

# ClinicalTrials.gov Identifier

NCT06229444

## **Document Name**

Data Use and Permissions Agreement (DUPA)\_v1.2

**Document Date** 

February 8, 2024

## **Predict + Protect Data Use and Permissions Agreement (DUPA)**

TITLE: Predict + Protect: A randomized controlled trial exploring the

effectiveness of a predictive health education intervention on the adoption of protective behaviors related to influenza-like illness

(ILI)

PROTOCOL NO.: NA

WCG IRB Protocol #20240213

**SPONSOR:** Evidation Health, Inc.

**INVESTIGATOR:** Ernesto Ramirez, PhD, BS, MS

63 Bovet Rd #146

San Mateo, California 94402

**United States** 

HELP & SUPPORT help@evidation.com

**CONTACT INFORMATION:** 1 (650) 897-5968 (Voicemail available 24 hours)

Taking part in this survey is voluntary. You may decide not to participate, or you may leave the survey at any time. Your decision will not result in any penalty or loss of benefits to which you are otherwise entitled.

If you have any questions, concerns, or complaints or think this activity has hurt you, talk to the team at the phone number(s) listed in this document.

Thank you for your interest in this survey supported by Evidation. We'd like to ask you some questions about your thoughts and/or experiences related to staying healthy during the flu and cold season. In this survey, please think about your experiences with the following respiratory viral illnesses: flu, respiratory syncytial virus (RSV), and/or COVID-19.

#### What do I have to do to participate, and how long will this take?

To participate, you must choose "Yes" below and complete this survey. It should take about {xx} minutes to complete.

You may also receive additional surveys related to your experiences with the following respiratory viral illnesses in the future. Each time you will be provided this information and be asked to participate.

## What if I don't want to participate or stop participating? What other choices do I have?

You can choose to stop participating at any time by closing the survey, or clicking "Done" in the top right corner. If you have already started the survey, any answers you have provided may be saved and used for the objectives outlined above.

If you do not want to participate you may choose to close this survey now or respond "No" below.

#### What happens to me if I agree to participate in this survey?

If you decide to complete the survey, we will analyze your responses combined with additional information you've contributed in the past, and information you contribute in the future related to staying healthy during the cold and flu season. We will also share your coded data (meaning that your directly identifying information is removed and replaced with a code) with external research partners (such as government institutions and their partners, pharmaceutical companies, and other external research collaborators).

#### Will I be compensated for participating?

Yes, you will earn {xx} Evidation points for agreeing to participate and completing this survey.

## Is there any benefit to participating in this survey?

It is not expected you will personally benefit from participating. However, we will work with our partners to better understand experiences related to respiratory viruses. If you take part in this survey, the results may contribute to public health and scientific efforts related to respiratory viruses.

## Is there any risk to participating in this survey?

This is a minimal risk survey, which means that the risk of experiencing any harm or discomfort in this survey is not greater than the risk you would encounter in daily life. You will not receive any treatment as part of this survey. There are potential privacy and security risks that your survey information could be subject to unauthorized access or your data could be linked to you.

## What data may be collected from me or analyzed as part of this project?

- Click 'Yes' below to give us permission to combine your answers from this survey with the following information you've already contributed, and continue to contribute, as you use the Evidation platform. This includes the following data (when available).
  - Self-reported demographic information such as:
    - Age
    - Height
    - Weight
    - Birth Sex
    - Gender
    - Race/Ethnicity

- Education Status
- Employment Status
- Caregiver Status
- Household Size
- Relationship Status
- Household Income
- Health Insurance Type
- Zip Code
- Self-reported information about your health conditions such as:
  - Condition diagnosis
  - Treatment experience
  - Medical Care experience
  - Self-reported lab values
  - Condition Symptoms
  - Well-being and Quality of Life
- o Daily check-ins
  - Mood
  - Sleep quality
  - Quality of life
- O Responses to surveys you complete about your thoughts and/or experiences related to staying healthy during the cold and flu season (including experience with flu-like symptoms and illnesses) between {study start and end dates}.
- O All of your available activity data collected from {"Launch 90 days" to "launch + 5 months"} from connected devices you have linked to your Evidation account, as described below. For example:
  - Physical activity (for example, steps, wheelchair pushes, workouts, energy or calories burned)
  - Sleep performance (for example, duration, stages, disturbances, latency, overall quality)
  - Heart rate and heart rate variability (if available)
  - Body temperature (if available)
  - Oxygen saturation (if available)
  - Respiratory rate (if available)
  - Stand time (if available)
  - Physical capacity (for example, VO2 max; if available)
  - Stress (if available)

## Who will have access to my data and how will it be used?

Limited Evidation team members will have access to the coded dataset (meaning that your directly identifying information is removed and replaced with a code) created from your completion of the one-time survey and other permissioned data described above in order to conduct an analysis.

We may share some or all of the coded dataset and analysis of the aggregated data with external research partners (such as government institutions and their partners, pharmaceutical companies, and other external research collaborators). We may also share the aggregated data and analysis of the aggregated data on our blog, on a public site, with potential sponsors or partners, or in research publications. We will not share your directly identifying information (including your name or contact information) without your express permission. Your responses to the survey will be retained by us and may be used to help match you with future research or related opportunities where you can contribute and earn rewards. If you choose to delete your Evidation account, any coded data that has been archived as part of the analysis will not be subject to data deletion requests, and any previous coded data sharing with external research partners before receiving the data deletion request cannot be reversed.

## What if I have questions?

If you have any questions about this survey, please contact us at <a href="mailto:help@evidation.com">help@evidation.com</a> or submit a support request.

Responses to this survey are subject to our <u>Privacy Notice</u> and <u>Terms of Use</u>.

This research is being overseen by WCG IRB. An IRB is a group of people who perform independent review of research studies. You may talk to them at 855-818-2289 or clientcare@wcgclinical.com if:

- You have questions, concerns, or complaints that are not being answered by the research team
- You are not getting answers from the research team.
- You cannot reach the research team.
- You want to talk to someone else about the research.
- You have questions about your rights as a research subject.
- 1. Do you wish to complete this survey and share your information as outlined above?
  - a. Yes
  - b. No